CLINICAL TRIAL: NCT04264806
Title: A Phase 2, Randomized, Open-label Study of Cusatuzumab in Combination With Azacitidine Compared With Azacitidine Alone in Patients With Higher-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) and Who Are Not Candidates for Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: A Study of Cusatuzumab in Combination With Azacitidine Compared With Azacitidine Alone in Patients With Higher-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) and Who Are Not Candidates for Hematopoietic Stem Cell Transplantation (HSCT)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The cusatuzumab MDS strategy is under revision
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108734; 2019-003576-40 (EudraCT Number); 74494550MDS2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacitidine: Participants with MDS or CMML (Experimental): Participants with higher-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) will receive azacitidine 75 milligram per meter square (mg/m^2) body surface area (BSA) subcutaneously or Intravenously per local label on Days 1 through Day 7 of each 28-day cycle. Participants will be treated until disease progression; relapse from complete remission (CR), partial remission (PR), or marrow complete remission (mCR); transformation to acute myeloid leukemia (AML); death; or unacceptable toxicity.
  Interventions: Drug: Azacitidine
- Azacitidine and Cusatuzumab: Participants with MDS or CMML (Experimental): Participants with higher-risk MDS or CMML will receive azacitidine 75 mg/m^2 BSA subcutaneously or Intravenously per local label on Days 1 through 7 and cusatuzumab 20 mg/kg IV on Days 3 and 17 of each 28-day cycle. Participants will be treated until disease progression; relapse from CR, PR, mCR; transformation to AML; death; or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Cusatuzumab

INTERVENTIONS:
Drug: Azacitidine — Participants will receive subcutaneous (SC) or intravenous (IV) injection of Azacitidine 75 mg/m^2.
Drug: Cusatuzumab — Participants will receive SC or IV injection of Cusatuzumab 20 mg/kg.
  Other Names: JNJ-74494550,; ARGX-110
  Arms: Azacitidine and Cusatuzumab: Participants with MDS or CMML

SUMMARY:
The purpose of the study is to compare overall response rate (ORR) between treatment groups in participants with higher-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) who are not eligible for Hematopoietic Stem Cell Transplantation (HSCT).

DETAILED DESCRIPTION:
Cusatuzumab (also known as JNJ-74494550 and ARGX-110) is a humanized monoclonal antibody of camelid origin that binds with high affinity to human Cluster of Differentiation 70 (CD70). Azacitidine (an Hypomethylating agent [HMA]) is approved for the treatment of higher-risk MDS in the United States (US) and the European Union (EU). Both approvals are based on data showing decreased transfusion burden, delayed progression to acute myeloid leukemia (AML), improved quality of life, and extended survival. It is hypothesized that the addition of cusatuzumab to azacitidine will result in an improvement in overall response rate (ORR) compared with azacitidine alone in participants with higher-risk MDS or CMML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of de novo or secondary higher-risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) per World Health Organization (WHO) 2016 criteria
* At study entry, higher-risk MDS (intermediate, high, and very high risk MDS per Revised International Prognostic Scoring System [IPSS R]) OR higher-risk CMML (intermediate-2 or high risk CMML per CMML-specific Prognostic Scoring System [CPSS-Mol]). Participants with previous lower-risk MDS or CMML that has evolved to higher-risk MDS or CMML are eligible
* At study entry, not a candidate for Hematopoietic Stem Cell Transplantation (HSCT)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Adequate liver and renal function defined as follows: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) less than (<) 3 * upper limit of normal (ULN); Total bilirubin less than or equal to (<=) 1.5 * ULN, unless bilirubin rise is due to Gilbert's syndrome or of non hepatic origin; and Creatinine clearance (CrCl) greater than (>) 30 milliliter per minute per 1.73 square meters (mL/min/1.73 m^2) (by Modification of Diet in Renal Disease formula)

Exclusion Criteria:

* Received prior HSCT or any prior treatment, including hypomethylating agent (HMAs), for higher-risk MDS or CMML. Prior supportive therapies including transfusion and growth factors are acceptable
* Received prior treatment with cusatuzumab
* Presence of the breakpoint cluster region protein-Abelson murine leukemia (bcr-abl) rearrangement
* Received a live, attenuated vaccine within 4 weeks prior to initiation of study drug
* Any active systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2022-04-19 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 4 years
  ORR is a composite of complete remission (CR), partial remission (PR) and marrow complete remission (mCR) as per modified International Working Group (IWG) criteria.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Complete Remission (CR) | Up to 4 years
  Percentage of participants achieving CR as per IWG criteria will be reported.
Percentage of Participants who Achieve Transfusion Independence | Up to 4 years
  Percentage of participants who achieve transfusion independence will be reported. Transfusion independence is defined as a period of greater than or equal to (>=) 56 consecutive days with no transfusion occurring between the first and last dose of study drug +30 days.
Time to Transformation of Participants to Acute Myeloid Leukemia (AML) | Up to 4 years
  Time to transformation of participants to AML will be reported. Transformation to AML is defined as >= 20% bone marrow blasts.
Progression Free Survival (PFS) | Up to 4 years
  PFS is defined as the time from randomization to disease progression; relapse from CR, PR, or mCR; or death from any cause.
Overall Survival (OS) | Up to 4 years
  OS is defined as the time from randomization to death.
Hematologic Improvement Rate | Up to 4 years
  Hematologic improvement rate is defined as erythroid response (pretreatment, less than (<) 11 g/dL; hemoglobin >= 1.5 g/dL; relevant reduction of units of RBC transfusions by an absolute number of >= 4 Red blood cell (RBC) transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a hemoglobin of <= 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation; platelet response (pretreatment <100*10^9/L); absolute increase of >= 30*109/L for participants starting with >20*10^9/L platelets; increase to >20*109/L and by >= 100% for participants starting with <= 20*109/L platelets; Neutrophil response (pretreatment <1.0×10^9/L); and at least 100% increase and an absolute increase of >0.5*10^9/L.
Percentage of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 4 years
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Percentage of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Up to 4 years
  Percentage of participants with clinically significant abnormalities in laboratory parameters will be reported.
Area Under the Serum Concentration-Time Curve Within Timespan t1 to t2 (AUC[t1-t2]) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  The AUC(t1-t2) is the area under the serum concentration-time curve within timespan t1 to t2.
Maximum Serum Concentration (Cmax) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  Cmax is the maximum observed serum concentration.
Minimum Serum Concentration (Cmin) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  Cmin is the minimum observed serum concentration.
Elimination Half-Life (t1/2) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  T1/2 is the time measured for the serum concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Systemic Clearance (CL) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of Distribution (Vz) of Cusatuzumab | Cycle 1: Day 3,17 (predose, end of infusion [EOI] postdose), Day 4 (24 hours postdose) Cycle 2, 3, 4, 8, 11: Day 3 (predose, EOI postdose); Cycle 4 Day 21 to Cycle 5: Day 1(at disease evaluation); and end of treatment (EOT) [up to 4 years])
  The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Number of Participants with Developed Antidrug Antibodies to Cusatuzumab | Cycle 1: Day 3 (Predose); Cycle 1: Day 17 (Predose); Cycle 2: Day 3 (Predose); Cycle 8 and 11: Day 3 (Predose) and EOT (up to 4 years)
  Venous blood samples are analyzed for presence of antidrug antibodies to cusatuzumab. Participants with titer of confirmed positive samples for cusatuzumab antibodies are reported.
Percentage of Participants Achieving Complete Remission (CR) and Partial Remission (PR) | Up to 4 years
  Percentage of participants achieving CR and PR as per IWG criteria will be reported.
Time to response | Up to 4 years
  Time to response for participants who achieved CR, PR and mCR responses, defined as time from randomization to achieving the first response of CR, PR, or mCR as per modified IWG criteria.
Duration of response | Up to 4 years
  Time from achieving the first response of CR, PR, or mCR to relapse or death from any cause for those participants who responded.
Percentage of Participants With Clinically Meaningful Improvement in Functional Assessment of Cancer Therapy - Anemia Trial Outcome Index (FACT-An TOI) Total Score | Up to 4 years
  FACT-An is a scale in Functional Assessment of Chronic Illness Therapy Measurement System. It consists of Functional Assessment of Cancer Therapy (general version; FACT-G) and 20 questions labeled "additional concerns" that measure anemia/fatigue. FACT-G is 27-item compilation of general questions divided into 4 primary quality of life domains: physical well-being, social/family well-being, emotional wellbeing, and functional well-being. Participants will be asked to rate scale items as it applies to past 7 days, on 5-point scale (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). Negatively stated items will be reversed by subtracting the response from 4. After reversing the proper items, items are summed to a total to generate a score on (sub)scale. A summary Trial Outcome Index total score (FACT An TOI) will be calculated by summing physical well being, functional well being, and anemia symptoms subscales and higher is the score better is the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trials, Study Director — Janssen Research & Development, LLC
Locations (73):
- Australia (6):
  - St Vincents Hospital Sydney, Darlinghurst
  - St Vincents Hospital Melbourne, Fitzroy
  - Peter MacCallum Cancer Institute, Melbourne
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
  - Wollongong Hospital, Wollongong
- Brazil (9):
  - Hospital Erasto Gaertner- Liga Paranaense de Combate ao Câncer, Curitiba
  - Cepon - Centro De Pesquisas Oncologicas, Florianópolis
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto do cancer -COR -Hospital Mae de Deus, Porto Alegre
  - Oncoclínicas, Rio de Janeiro
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto
  - Hospital Paulistano, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
- France (9):
  - CHU d'Angers, Angers
  - Hopital Saint Vincent de Paul, Lille
  - CHU de Limoges, Hopital Dupuytren, Limoges
  - Hôpital de La Conception, Marseille
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint-Louis, Paris
  - Hopital Cochin APHP, Paris
  - CHRU Tours Hôpital Bretonneau, Tours
  - CHU de Nancy_ Hôpital Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar an der Technischen Universität München, München
  - Universitaetsklinikum Ulm, Ulm
- Italy (8):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria di Ferrara, Cona
  - Università del Piemonte Orientale - Ospedale Maggiore della Carità di Novara, Novara
  - Aou San Luigi Gonzaga, Orbassano
  - Grande Ospedale Metropolitano 'Bianchi-Melacrino-Morelli' Reggio Calabria, Reggio Calabria
  - Fondazione Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - Istituto Clinico Humanitas, Rozzano
- Russia (8):
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - Saint Petersburg City Hospital #15, Saint Petersburg
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - St.-Petersburg City Clinical Hospital nr 31, Saint Petersburg
  - Oncology Dispensary of Komi Republic, Syktyvkar
- Saudi Arabia (3):
  - King Fahad Specialist hospital, Dammam
  - King Abdulaziz Medical City, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Spain (9):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. Univ. Infanta Leonor, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hosp. Univ. Son Espases, Palma
  - Hosp. Clinico Univ. de Salamanca, Salamanca
  - Hosp. Virgen Del Rocio, Seville
- Switzerland (3):
  - INSELSPITAL, Universitätsspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - UniversitaetsSpital Zuerich, Zurich
- Turkey (Türkiye) (7):
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Koc Universitesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
- United Kingdom (5):
  - St James Hospital, Leeds
  - University College London Hospitals, London
  - Kings College Hospital, London
  - Royal Victoria Infirmary, Newcastle Upun Tyne
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency